CLINICAL TRIAL: NCT01034605
Title: The Effect of PinnoThin on Satiety and Food Intake
Acronym: PinnoThin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HumBio_Westerterp08
Record Dates: First submitted 2009-12-02; First posted 2009-12-17 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- inulin (Experimental): oligofructose
  Interventions: Dietary Supplement: PinnoThin

INTERVENTIONS:
Dietary Supplement: PinnoThin — 6.0 gram of the oil extract from the korean pine nut (PinnoThin) as a single dose

SUMMARY:
Based upon an increased secretion of gastrointestinal satiety hormones (CCK, GLP-1), PinnoThin is hypothesized to be more satiating, and to limit energy intake in humans. Therefore, the objective of this study is to investigate whether PinnoThin leads to an increase in satiety as determined by VAS ratings? Additionally, does PinnoThin consumed during breakfast, in comparison to placebo, in overweight women, lead to a decrease in energy intake during an ad libitum lunch?

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and under 45
* women
* BMI over 23 and under 30
* breakfast eaters

Exclusion Criteria:

* men
* age under 18 and over 45
* BMI under 23 and over 30
* use of medication
* pregnant and breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
appetite profile ratings | 10 timepoints

SECONDARY OUTCOMES:
energy intake | 3.5 hours after PinnoThin

CONTACTS AND LOCATIONS:
Overall Officials: Klaas R Westerterp, Prof, Principal Investigator — NUTRIM
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Verhoef SP, Westerterp KR. No effects of Korean pine nut triacylglycerol on satiety and energy intake. Nutr Metab (Lond). 2011 Nov 10;8(1):79. doi: 10.1186/1743-7075-8-79. PMID 22074178